CLINICAL TRIAL: NCT06711120
Title: Randomized Controlled Study of Radio Frequency and Microwave of the Small Saphenous Vein
Brief Title: Comparative Analysis of Radiofrequency Ablation and Microwave Ablation Procedures for the Treatment of Small Saphenous Varicose Veins
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chengdu University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Chunshui He, chief physician, Chengdu University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ChengduUTCMvs8
Record Dates: First submitted 2024-11-17; First posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Varicose Veins of Lower Limb; Venous Insufficiency of Leg; Vascular Disease，Peripheral
Keywords: varicose veins of the small saphenous veins; radiofrequency ablation; microwave ablation
MeSH Terms: conditions — Peripheral Vascular Diseases | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiofrequency ablation for the treatment of varicose veins of the small saphenous vein (Experimental): After radiofrequency ablation, patients' postoperative length of stay, time out of bed, and visual analogue scoring (VAS) scores were used to count the occurrence of postoperative complications, and all patients were followed up with colour Doppler ultrasound at 2 weeks, 1 month, and 3 months postoperatively to determine whether there was recurrence or not, and the use of the Venous Clinical Criticality Score (VCSS), Aberdeen Varicose Vein Questionnaire (AVVQ), and Chronic Venous Disease Quality of Life Scale (CIVIQ) to evaluate the treatment effect.
  Interventions: Procedure: Radiofrequency ablation and microwave ablation are used to treat small saphenous varicose veins, respectively
- Microwave ablation for the treatment of varicose veins of the small saphenous vein (Experimental): After Microwave ablation, patients' postoperative length of stay, time out of bed, and visual analogue scoring (VAS) scores were used to count the occurrence of postoperative complications, and all patients were followed up with colour Doppler ultrasound at 2 weeks, 1 month, and 3 months postoperatively to determine whether there was recurrence or not, and the use of the Venous Clinical Criticality Score (VCSS), Aberdeen Varicose Vein Questionnaire (AVVQ), and Chronic Venous Disease Quality of Life Scale (CIVIQ) to evaluate the treatment effect.
  Interventions: Procedure: Radiofrequency ablation and microwave ablation are used to treat small saphenous varicose veins, respectively

INTERVENTIONS:
Procedure: Radiofrequency ablation and microwave ablation are used to treat small saphenous varicose veins, respectively — During the procedure, 2% lidocaine was injected subcutaneously along the course of the saphenous vein under ultrasound guidance, and after local anaesthesia, an incision was made at the ankle joint of the saphenous vein to locate the saphenous vein, and a radiofrequency guidewire and catheter sheath were introduced.The saphenous vein was incised at the ankle joint under local anaesthesia. Under ultrasound monitoring, the radiofrequency catheter was placed in the saphenous popliteal vein at a distance of 1~2 cm and the position of the catheter was fixed, and then anaesthesia and swelling fluid was injected into the fascial tissues around the main trunk of the small saphenous vein in segments.The two groups were treated with radiofrequency ablation and microwave ablation surgery, respectively.

SUMMARY:
Objective: To investigate the clinical efficacy of ultrasound-guided radiofrequency ablation and microwave ablation in the treatment of primary saphenous varicose veins.

DETAILED DESCRIPTION:
Chronic venous insufficiency (CVI) is a common clinical disease, and varicose veins of the lower extremities are the main clinical manifestations of CVI, and studies have shown that the prevalence of CVI is 10%~25%.Although small saphenous varicose veins are rare, accounting for only 15% of great saphenous varicose veins, the surgical treatment of small saphenous varicose veins is more challenging due to the small saphenous varicose veins injected into the popliteal vein.In the late 19th and early 20th centuries, high ligation was the only treatment for the small saphenous varicose veins, however, it had a high recurrence rate and increased risk of nerve injury due to the presence of the small saphenous vein with the sural nerve. In open surgery for small saphenous varicose veins, about 26% of patients can be complicated by sural neuropathy, and due to changes in their anatomy, about 22% of patients do not adequately identify the proximal saphenous vein or saphenopopliteal fossa junction intraoperatively, even if the location is determined by ultrasound preoperatively.Since conventional surgery is more traumatic and has more complications, it is not favorable to the patient's postoperative recovery. In recent years, with the development of venous vascular ultrasound imaging technology, ultrasound-guided radiofrequency ablation and microwave ablation have gradually been widely used in the treatment of small saphenous varicose veins. Compared with conventional surgical procedures, radiofrequency ablation and microwave ablation are less invasive, safer and more effective for saphenous varicose veins, but not many studies have been conducted on the safety and efficacy of small saphenous varicose veins. Therefore, the aim of this study was to investigate the clinical efficacy of ultrasound-guided radiofrequency ablation versus microwave ablation in the treatment of primary small saphenous varicose veins.Translated with DeepL.com (free version)

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years and ≤90 years;
* Clinical diagnosis of primary varicose veins of the lower extremities, CEAP clinical classification C2-C6, requiring treatment of the great and/or small saphenous vein segments, and at least 1 of the clinical symptoms of swelling, pain, burning sensation, heaviness, easy fatigue, itchy skin, and night cramps;
* Valve insufficiency of the great saphenous vein, small saphenous vein, or transport vein;
* Doppler ultrasound confirmation of a saphenous vein diameter greater than 3 mm and less than 12 mm in the standing position;
* Only one limb per patient was selected for inclusion in the study;
* Patients signed an informed consent form and were willing to co-operate in completing the protocol-specified investigations and follow-up visits.

Exclusion Criteria:

* Thrombosis of the great saphenous or small saphenous vein, or combined deep vein thrombosis, or previous history of deep vein thrombosis or pulmonary embolism.
* Recurrent varicose veins after previous treatment.
* Severe distortion of the great saphenous vein with anticipated catheter failure.
* Severe lower limb ischaemia (CLI) (ABPI <0.8).
* Known allergy to medications and device materials involved in the study.
* Pre-existing implanted pacemaker, defibrillator, currently on regular anticoagulation therapy (e.g., warfarin, heparin).
* Women who are pregnant or breastfeeding.
* Unable or unwilling to complete the questionnaire.
* Participating in a study of another drug or device.
* Life expectancy <1 year.
* Those undergoing treatment for skin malignancies other than non-melanoma.
* Daily use of narcotic drugs or non-steroidal anti-inflammatory drugs to control pain due to venous disease.
* In the judgement of the investigator, endovenous therapy is not appropriate.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
6-month postoperative occlusion rate | 6 months after surgery
  occlusion defined as no flow recirculation of the closed treated segment of the vein as confirmed by Doppler ultrasound

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of Chengdu University of Traditional Chinese Medicine, Chengdu, China

IPD SHARING:
Plan to Share IPD: No